CLINICAL TRIAL: NCT05707767
Title: A Prospective Study of Surgical Treatment Strategies for Chordoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XW-NS-CHORC
Record Dates: First submitted 2022-10-09; First posted 2023-02-01 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-10

CONDITIONS: Chordoma of Spine; Surgery
Keywords: chordoma
MeSH Terms: conditions — Chordoma | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chordoma Patients (Experimental): Chordoma Patients
  Interventions: Procedure: Resection surgery

INTERVENTIONS:
Procedure: Resection surgery — Patients undergo resection surgery in our hospital.

SUMMARY:
Chordoma is a rare but locally invasive cancer that arises from the embryonic notochord. Total resection is challenging in mobile spine because of the complex anatomy and bone invasion.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 70 ys,
* With a diagnosis of chordoma confirmed by pathology,
* Undergone surgical treatment in our hospital,
* Available for clinical follow-up and agree to long-term clinical follow-up and sign informed consent.

Exclusion Criteria:

* Suffer from other tumors,
* Suffer from cardiovascular disease, cerebrovascular disease, or immune system disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Excision Extension | 1 week after surgery.
  Clinical and radiographic assessments of excision extension of tumor.

SECONDARY OUTCOMES:
OS (Overall Survival) | 2 years
  Overall Survival of patient underwent surgery.
PFS (Progression-Free Survival) | 2 years
  Progression-Free Survival of patient underwent surgery.
DFS (Disease Free Survival) | 2 years
  Disease Free Survival of patient underwent surgery.
ORR (Objective Response Rate) | 2 years
  Objective Response Rate of patient underwent surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Result] Walcott BP, Nahed BV, Mohyeldin A, Coumans JV, Kahle KT, Ferreira MJ. Chordoma: current concepts, management, and future directions. Lancet Oncol. 2012 Feb;13(2):e69-76. doi: 10.1016/S1470-2045(11)70337-0. PMID 22300861
- [Result] Wedekind MF, Widemann BC, Cote G. Chordoma: Current status, problems, and future directions. Curr Probl Cancer. 2021 Aug;45(4):100771. doi: 10.1016/j.currproblcancer.2021.100771. Epub 2021 Jul 1. PMID 34266694
- [Result] Yeter HG, Kosemehmetoglu K, Soylemezoglu F. Poorly differentiated chordoma: review of 53 cases. APMIS. 2019 Sep;127(9):607-615. doi: 10.1111/apm.12978. PMID 31243811
- [Result] Kolz JM, Wellings EP, Houdek MT, Clarke MJ, Yaszemski MJ, Rose PS. Surgical treatment of primary mobile spine chordoma. J Surg Oncol. 2021 Apr;123(5):1284-1291. doi: 10.1002/jso.26423. Epub 2021 Feb 10. PMID 33567141
- [Result] Williams BJ, Raper DM, Godbout E, Bourne TD, Prevedello DM, Kassam AB, Park DM. Diagnosis and treatment of chordoma. J Natl Compr Canc Netw. 2013 Jun 1;11(6):726-31. doi: 10.6004/jnccn.2013.0089. PMID 23744869